CLINICAL TRIAL: NCT03770910
Title: The Effect of GIP(3-30)NH2
Acronym: GA-10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Lærke Smidt Gasbjerg, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SDCC_CMP_GA-10
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Endocrine - Other
Keywords: GIP; Insulin secretin; Incretin hormone
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo+placebo (Placebo Comparator): Saline infusions
  Interventions: Other: Saline
- GIP+placebo (Active Comparator): GIP(1-42), receptor agonist
  Interventions: Other: GIP receptor agonist; Other: Saline
- GIP+dose 1 (Experimental): GIP(1-42) and lowest dose of GIP(3-30)NH2
  Interventions: Other: GIP receptor antagonist; Other: GIP receptor agonist
- GIP+dose 2 (Experimental): GIP(1-42) and dose of GIP(3-30)NH2
  Interventions: Other: GIP receptor antagonist; Other: GIP receptor agonist
- GIP+dose 3 (Experimental): GIP(1-42) and dose of GIP(3-30)NH2
  Interventions: Other: GIP receptor antagonist; Other: GIP receptor agonist
- GIP+dose4 (Experimental): GIP(1-42) and highest dose of GIP(3-30)NH2
  Interventions: Other: GIP receptor antagonist; Other: GIP receptor agonist

INTERVENTIONS:
Other: GIP receptor antagonist — GIP receptor antagonist
  Arms: GIP+dose 1; GIP+dose 2; GIP+dose 3; GIP+dose4
Other: GIP receptor agonist — GIP(1-42)
  Arms: GIP+dose 1; GIP+dose 2; GIP+dose 3; GIP+dose4; GIP+placebo
Other: Saline — Placebo (vehicle for infusions)
  Arms: GIP+placebo; Placebo+placebo

SUMMARY:
Infusion of glucose-dependent insulintropic polypeptide (GIP) receptor antagonist and evaluation of effect of insulin secretion in healthy subjects.

DETAILED DESCRIPTION:
Infusion of glucose-dependent insulintropic polypeptide (GIP) receptor antagonist and evaluation of effect of insulin secretion in healthy subjects.

Six study hyperglycemic clamps (10 mmol/l) pr. participant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI 19-28 kg/m*m
* Stable body weight

Exclusion Criteria:

* Diabetes
* Anemia
* First-degree relatives with diabetes

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Insulin secretion | 8 weeks
  Insulin secretion rates (ISR) calculated from serum levels of C-peptide

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Clinical Metabolic Physiology, Gentofte Municipality, Copenhagen
  - Clinical Metabolic Physiology, Copenhagen, Gentofte

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers unless data management agreements are signed.